CLINICAL TRIAL: NCT01004614
Title: An Open, Randomized, Parallel-Cohort, 2-Periods, Crossover, Single Dose Bioequivalence Study For 5 Mg Amlodipine Orally-Disintegrating Tablet In Healthy Male Subjects
Brief Title: Bioequivalence Study For 5 Mg Amlodipine Orally-Disintegrating Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A0531088
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Results first posted 2012-01-04 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Healthy
MeSH Terms: interventions — Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): 24 subjects (12 subjects per sequence) will receive treatment A) one 5 mg amlodipine 3rd OD tablet (test) with water and treatment B) one 5 mg amlodipine 2nd OD tablet (reference) with water.
  Interventions: Drug: Amlodipine
- Cohort 2 (Active Comparator): 24 subjects (12 subjects per sequence) will receive treatment C) one 5 mg amlodipine 3rd OD tablet (test) without water, and treatment D) one 5 mg amlodipine 2nd OD tablet (reference) without water
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Amlodipine — 3rd OD 5 mg tablet single oral dose administered with water
  Arms: Cohort 1
Drug: Amlodipine — 2nd OD 5 mg tablet single oral dose administered with water
  Arms: Cohort 1
Drug: Amlodipine — 3rd OD 5 mg tablet single oral dose administered without water
  Arms: Cohort 2
Drug: Amlodipine — 2nd OD 5 mg tablet single oral dose administered without water
  Arms: Cohort 2

SUMMARY:
This study is being conducted to determine if 5 mg amlodipine 3rd Orally-Disintegrating (OD) tablet (new formulation) and 5 mg amlodipine 2nd OD tablet (commercial formulation) are bioequivalent.

ELIGIBILITY:
Inclusion Criteria:

* Healthy;
* Body Mass Index (BMI) of 18 to 28 kg/m2;
* total body weight within the range of 50 to 100 kg

Exclusion Criteria:

* History of regular alcohol consumption exceeding 14 drinks/week
* Use of tobacco- or nicotine-containing products in excess of the equivalent of 10 cigarettes per day

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Minato-ku, Tokyo, Japan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0531088&StudyName=Bioequivalence%20Study%20For%205%20Mg%20Amlodipine%20Orally-Disintegrating%20Tablet

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened at one center in Japan.
Pre-assignment Details: This study consisted of 2 cohorts (I and II). The design of each cohort was an open-label, randomized, 2-periods, crossover, single-dose study in healthy adult male subjects. A washout period of at least 14 days was taken between each administration in Periods 1 and 2.
Groups:
- 3rd OD Tablet With Water, Then 2nd OD Tablet With Water: One amlodipine third generation orally disintegrating (OD) 5 mg tablet (test) taken with water during the first intervention period, then one amlodipine second generation OD 5 mg tablet (reference) taken with water during second intervention period. A washout of 14 days was retained between periods.
- 2nd OD Tablet With Water, Then 3rd OD Tablet With Water: One amlodipine second generation OD 5 mg tablet (reference) taken with water during the first intervention period, then one amlodipine third generation OD 5 mg tablet (test) taken with water during the second intervention period. A washout of 14 days was retained between periods.
- 3rd OD Tablet Without Water, Then 2nd OD Tablet Without Water: One amlodipine third generation OD 5 mg tablet (test) taken without water during the first intervention period, then one amlodipine second generation OD 5 mg tablet (reference) taken without water during the second intervention period. A washout of 14 days was retained between periods.
- 2nd OD Tablet Without Water, Then 3rd OD Tablet Without Water: One amlodipine second generation OD 5mg tablet (reference) taken without water during the first intervention period, then one amlodipine third generation OD 5 mg tablet (test) taken without water during the second intervention period. A washout of 14 days was retained between periods.
Period: First Intervention
Arm/Group | 3rd OD Tablet With Water, Then 2nd OD Tablet With Water | 2nd OD Tablet With Water, Then 3rd OD Tablet With Water | 3rd OD Tablet Without Water, Then 2nd OD Tablet Without Water | 2nd OD Tablet Without Water, Then 3rd OD Tablet Without Water
Started | 12 | 12 | 12 | 12
Completed | 12 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0
Period: Washout
Arm/Group | 3rd OD Tablet With Water, Then 2nd OD Tablet With Water | 2nd OD Tablet With Water, Then 3rd OD Tablet With Water | 3rd OD Tablet Without Water, Then 2nd OD Tablet Without Water | 2nd OD Tablet Without Water, Then 3rd OD Tablet Without Water
Started | 12 | 12 | 12 | 12
Completed | 12 | 11 | 12 | 12
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Second Intervention
Arm/Group | 3rd OD Tablet With Water, Then 2nd OD Tablet With Water | 2nd OD Tablet With Water, Then 3rd OD Tablet With Water | 3rd OD Tablet Without Water, Then 2nd OD Tablet Without Water | 2nd OD Tablet Without Water, Then 3rd OD Tablet Without Water
Started | 12 | 11 | 12 | 12
Completed | 12 | 11 | 12 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 3rd OD Tablet With Water, Then 2nd OD Tablet With Water: One amlodipine third generation orally disintegrating (OD) 5 mg tablet (test) taken with water during the first intervention period, then one amlodipine second generation OD 5 mg tablet (reference) taken with water during the second intervention period. A washout of 14 days was retained between periods.
- 2nd OD Tablet With Water, Then 3rd OD Tablet With Water: One amlodipine second generation OD 5mg tablet (reference) taken with water during the first intervention period, then one amlodipine third generation OD 5 mg tablet (test) taken with water during the second intervention period. A washout of 14 days was retained between periods.
- Total: Total of all reporting groups
Arm/Group | 3rd OD Tablet With Water, Then 2nd OD Tablet With Water | 2nd OD Tablet With Water, Then 3rd OD Tablet With Water | 3rd OD Tablet Without Water, Then 2nd OD Tablet Without Water | 2nd OD Tablet Without Water, Then 3rd OD Tablet Without Water | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (10.7) | 32.4 (11.1) | 37.3 (9.0) | 37.8 (12.1) | 33.1 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 12 | 12 | 12 | 12 | 48

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-Time Curve From Zero Time Until the Last Sampling Time (AUCt)
Description: Area under the concentration-time curve from zero time until the last sampling time
Time Frame: prior to dosing, 2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120 and 144 hours post dose
Population: The PK parameter analysis set was defined as all subjects randomized and treated who completed the study.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Cohort I: 3rd OD Tablet (Test) With Water: Cohort I: One 5 mg amlodipine 3rd OD tablet (test) taken with water as a single oral dose
- Cohort I: 2nd OD Tablet (Reference) With Water: Cohort I: One 5 mg amlodipine 2nd OD tablet (reference) taken with water as a single oral dose
- Cohort II: 3rd OD Tablet (Test) Without Water: Cohort II: One 5 mg amlodipine 3rd OD tablet (test) taken without water as a single oral dose
- Cohort II: 2nd OD Tablet (Reference) Without Water: Cohort II: One 5 mg amlodipine 2nd OD tablet (reference) taken without water as a single oral dose
Arm/Group | Cohort I: 3rd OD Tablet (Test) With Water | Cohort I: 2nd OD Tablet (Reference) With Water | Cohort II: 3rd OD Tablet (Test) Without Water | Cohort II: 2nd OD Tablet (Reference) Without Water
Number analyzed (Participants) | 23 | 23 | 24 | 24
ng*h/mL | 126.36 (33.16) | 129.48 (39.93) | 122.33 (32.59) | 119.75 (28.23)
Statistical Analysis 1: Comparison: Cohort I: 3rd OD Tablet (Test) With Water vs Cohort I: 2nd OD Tablet (Reference) With Water vs Cohort II: 3rd OD Tablet (Test) Without Water vs Cohort II: 2nd OD Tablet (Reference) Without Water; Natural log transformed AUCt was analyzed using a mixed effects model with sequence, period and formulation as fixed effects and subject within sequence as a random effect. Adjusted mean difference (test - reference) and 90% CI was obtained from the model and exponentiated to provide estimates of the ratio of adjusted geometric mean and 90% CI for the ratio. Alternative hypothesis of bioequivalence: (H1: θL <=µT - µR <=θU); null hypothesis of inequivalence: (Ho: µT - µR <θL or µT - µR >θU); Test type: Non-Inferiority or Equivalence — Bioequivalence of the two formulations was concluded if the 90% confidence intervals for the ratio of adjusted geometric means for both AUCt and Cmax fell wholly within (80%, 125%); ratios of adjusted geometric mean = 98.61, 90% CI 2-sided [93.09 to 104.46] — Parameter estimate = ratio (%) (test/reference) of adjusted geometric means
Statistical Analysis 2: Comparison: Cohort I: 3rd OD Tablet (Test) With Water vs Cohort I: 2nd OD Tablet (Reference) With Water vs Cohort II: 3rd OD Tablet (Test) Without Water vs Cohort II: 2nd OD Tablet (Reference) Without Water; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratios of adjusted geometric mean = 101.29, 90% CI 2-sided [97.28 to 105.45] — Parameter estimate = ratio (%) (test/reference) of adjusted geometric means

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: prior to dosing, 2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120 and 144 hours post dose
Population: The PK parameter analysis set was defined as all subjects randomized and treated who completed the study.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort I: 3rd OD Tablet (Test) With Water | Cohort I: 2nd OD Tablet (Reference) With Water | Cohort II: 3rd OD Tablet (Test) Without Water | Cohort II: 2nd OD Tablet (Reference) Without Water
Number analyzed (Participants) | 23 | 23 | 24 | 24
ng/mL | 2.70 (0.513) | 2.74 (0.650) | 2.48 (0.470) | 2.45 (0.409)
Statistical Analysis 1: Comparison: Cohort I: 3rd OD Tablet (Test) With Water vs Cohort I: 2nd OD Tablet (Reference) With Water vs Cohort II: 3rd OD Tablet (Test) Without Water vs Cohort II: 2nd OD Tablet (Reference) Without Water; Natural log transformed Cmax was analyzed using a mixed effects model with sequence, period and formulation as fixed effects and subject within sequence as a random effect. Adjusted mean difference (test - reference) and 90% CI was obtained from the model and exponentiated to provide estimates of the ratio of adjusted geometric mean and 90% CI for the ratio. Alternative hypothesis of bioequivalence: (H1: θL <=µT - µR <=θU); null hypothesis of inequivalence: (Ho: µT - µR <θL or µT - µR >θU); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Parameter estimate = ratio (%) (test/reference) of adjusted geometric means; ratios of adjusted geometric mean = 99.30, 90% CI 2-sided [92.28 to 106.28]
Statistical Analysis 2: Comparison: Cohort I: 3rd OD Tablet (Test) With Water vs Cohort I: 2nd OD Tablet (Reference) With Water vs Cohort II: 3rd OD Tablet (Test) Without Water vs Cohort II: 2nd OD Tablet (Reference) Without Water; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Parameter estimate = ratio (%) (test/reference) of adjusted geometric means; ratios of adjusted geometric mean = 100.84, 90% CI 2-sided [95.93 to 106.00]

3. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUClast), Area Under the Plasma Concentration-Time Curve to Infinity (AUCinf)
Description: AUC last = Area under the concentration versus time curve from zero time until the last measurable concentration is calculated using the trapezoidal rule.
  AUCinf = AUClast + (Ct / kel), where Ct is the estimated concentration at the last measurable concentration.
Time Frame: prior to dosing, 2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120 and 144 hours post dose
Population: The PK parameter analysis set was defined as all subjects randomized and treated who completed the study.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort I: 3rd OD Tablet (Test) With Water | Cohort I: 2nd OD Tablet (Reference) With Water | Cohort II: 3rd OD Tablet (Test) Without Water | Cohort II: 2nd OD Tablet (Reference) Without Water
Number analyzed (Participants) | 23 | 23 | 24 | 24
ng*h/mL
  AUClast | 124.14 (33.96) | 127.36 (40.91) | 121.05 (33.76) | 118.27 (29.43)
  AUCinf | 142.87 (43.20) | 145.22 (49.19) | 140.41 (42.18) | 138.14 (34.10)

4. Secondary Outcome: Apparent Terminal Elimination Phase Rate Constant (Kel)
Description: Estimated as the absolute value of the slope of a linear regression during the terminal phase of the natural-logarithm (ln) transformed concentration-time profile.
Time Frame: prior to dosing, 2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120 and 144 hours post dose
Population: The PK parameter analysis set was defined as all subjects randomized and treated who completed the study.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Cohort I: 3rd OD Tablet (Test) With Water | Cohort I: 2nd OD Tablet (Reference) With Water | Cohort II: 3rd OD Tablet (Test) Without Water | Cohort II: 2nd OD Tablet (Reference) Without Water
Number analyzed (Participants) | 23 | 23 | 24 | 24
L/h | 0.0174 (0.0031) | 0.0179 (0.0035) | 0.0162 (0.0041) | 0.0156 (0.0031)

5. Secondary Outcome: Apparent Terminal Elimination Half-Life (T-half)
Description: Terminal phase half-life calculated as ln(2) / kel
Time Frame: prior to dosing, 2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120 and 144 hours post dose
Population: The PK parameter analysis set was defined as all subjects randomized and treated who completed the study.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Cohort I: 3rd OD Tablet (Test) With Water | Cohort I: 2nd OD Tablet (Reference) With Water | Cohort II: 3rd OD Tablet (Test) Without Water | Cohort II: 2nd OD Tablet (Reference) Without Water
Number analyzed (Participants) | 23 | 23 | 24 | 24
hour | 41.45 (9.76) | 40.27 (8.48) | 45.04 (10.16) | 46.20 (8.85)

6. Secondary Outcome: Mean Residence Time (MRT)
Description: MRT = AUMCinf / AUCinf, where AUMCinf is the area under the first moment curve from zero time to infinity calculated as AUMCinf = AUMCt + ((t x Ct) / kel) + (Ct / kel^2). AUMCt is the area under the first moment curve from zero time to time t calculated using the trapezoidal method.
Time Frame: prior to dosing, 2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120 and 144 hours post dose
Population: The PK parameter analysis set was defined as all subjects randomized and treated who completed the study.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Cohort I: 3rd OD Tablet (Test) With Water | Cohort I: 2nd OD Tablet (Reference) With Water | Cohort II: 3rd OD Tablet (Test) Without Water | Cohort II: 2nd OD Tablet (Reference) Without Water
Number analyzed (Participants) | 23 | 23 | 24 | 24
hour | 61.29 (13.55) | 59.77 (11.99) | 66.18 (14.10) | 67.33 (11.90)

7. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: prior to dosing, 2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120 and 144 hours post dose
Population: The PK parameter analysis set was defined as all subjects randomized and treated who completed the study.
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort I: 3rd OD Tablet (Test) With Water | Cohort I: 2nd OD Tablet (Reference) With Water | Cohort II: 3rd OD Tablet (Test) Without Water | Cohort II: 2nd OD Tablet (Reference) Without Water
Number analyzed (Participants) | 23 | 23 | 24 | 24
hour | 8 [4 to 12] | 8 [4 to 12] | 8 [6 to 12] | 8 [6 to 12]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Cohort I: 3rd OD Tablet (Test) With Water | Cohort I: 2nd OD Tablet (Reference) With Water | Cohort II: 3rd OD Tablet (Test) Without Water | Cohort II: 2nd OD Tablet (Reference) Without Water
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 7/23 | 6/24 | 2/24 | 3/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort I: 3rd OD Tablet (Test) With Water (N=23) | Cohort I: 2nd OD Tablet (Reference) With Water (N=24) | Cohort II: 3rd OD Tablet (Test) Without Water (N=24) | Cohort II: 2nd OD Tablet (Reference) Without Water (N=24)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Pharingitis (Infections and infestations) | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 1
Oropharyngeal disconfort (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.